CLINICAL TRIAL: NCT00830180
Title: PHASE 2 OPEN-LABEL SAFETY EXTENSION STUDY OF TANEZUMAB IN CANCER PATIENTS WITH PAIN DUE TO BONE METASTASES
Brief Title: Open Label Extension In Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A4091029; 2008-005182-66 (EudraCT Number); CANCER PAIN OL EXTENSION (Other: Alias Study Number)
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-02

CONDITIONS: Neoplasms; Bone Metastases
Keywords: Cancer pain; NGF; open-label extension
MeSH Terms: conditions — Neoplasms; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-NGF AB (Experimental)
  Interventions: Biological: Anti-NGF AB

INTERVENTIONS:
Biological: Anti-NGF AB — Solution for injection, 10 mg, one injection/8 weeks

SUMMARY:
To evaluate the safety and efficacy of anti-NGF AB in cancer patients with pain due to bone metastases who participated in the double-blind Study A4091003 and who wish to receive open-label therapy.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer, breast cancer, renal cell carcinoma or multiple myeloma that has been diagnosed as having metastasized to bone;
* Karnofsky Performance Score ≥40% at Baseline;
* patients randomized and treated with intravenous study drug in double-blind Study A4091003.

Exclusion Criteria:

* Patient was withdrawn from Study A4091003 for an adverse event or serious adverse event;
* Occurrence of any adverse event or condition during Study A4091003 or since termination from that study that, in the opinion of the Investigator, would put the patient at increased safety risk or should exclude the subject from participating in the open-label extension Study A4091029.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-10-29 (Actual); Primary Completion 2013-02-14 (Actual); Study Completion 2013-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (6):
  - UCSD Center for Pain Medicine, La Jolla, California
  - UCSD Medical Center - Thornton Hospital, La Jolla, California
  - UCSD Periman Ambulatory Care Center, La Jolla, California
  - UCSD Moores Cancer Center, La Jolla, California
  - WK River Cities Clinical Research Center, Shreveport, Louisiana
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Nuhr Zentrum, Senftenberg, Austria
- Clinic of Oncology, Banja Luka, Bosnia and Herzegovina
- General Hospital Varazdin, Varaždin, Croatia
- Fejer Megyei Szt. Gyorgy Korhaz - Rendelointezet/Aneszteziologiai es Intenziv Betegellato Osztaly, Székesfehérvár, Hungary
- India (3):
  - Central India Cancer Research Institute Central India Cancer Research Institute, Nagpur, Maharashtra
  - Shatabdi Super Speciality Hospital, Nashik, Maharashtra
  - Chhatrapati Shahuji Maharaj Medical University, Lucknow, Uttar Pradesh
- Latvian Oncology Centre, Riga, Latvia
- Poland (5):
  - Niepubliczny Zaklad Opieki Zdrowotnej, Bydgoszcz
  - Hospicjum im Ks Eugeniusza Dutkiewicza SAC w Gdansku, Gdansk
  - **Poradnia Medycyny Paliatywnej, Hospicjum Palium, Poznan
  - Wielkopolskie Centrum Onkologii im. Marii Sklodowskiej-Curie, Poznan
  - NZOZ Zespol Opieki Domowej Polskiego Towarzystwa Opieki Paliatywnej, Włocławek
- Slovakia (2):
  - Fakultna Nemocina s Poliklinikou FD Roosevelta Banska Bystrica, Banská Bystrica
  - Narodny onkologicky ustav, Bratislava
- South Korea (2):
  - Severance Hospital, Yonsei University College of Medicine, Seodaemun-gu, Seoul
  - Samsung Medical Center, Division of Hematology-Oncology, Department of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sopata M, Katz N, Carey W, Smith MD, Keller D, Verburg KM, West CR, Wolfram G, Brown MT. Efficacy and safety of tanezumab in the treatment of pain from bone metastases. Pain. 2015 Sep;156(9):1703-1713. doi: 10.1097/j.pain.0000000000000211. PMID 25919474
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091029&StudyName=Open%20Label%20Extension%20In%20Cancer%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Tanezumab 10 mg (A4091029): Participants received a single intravenous (IV) infusion of tanezumab 10 milligram (mg) administered at Visit 1 (Baseline, Day 1), Visit 4 (Day 57, Week 8), Visit 6 (Day 113, Week 16), and Visit 7 (Day 169, Week 24). For participants in Poland entering the Extended-use Period, tanezumab 10 mg was also administered via IV infusion at Visit 9 (Day 282, Week 40), Visit 10 (Day 337, Week 48), Visit 11 (Day 393, Week 56), and Visit 12 (Day 449, Week 64) with a plus or minus 5 day window for each post-baseline IV infusion.
Period: Overall Study
Arm/Group | Tanezumab 10 mg (A4091029)
Started | 41
Received Tanezumab in Parent Study A4091003 | 19
Received Placebo in Parent Study A4091003 | 22
Completed | 15
Not Completed | 26
Not completed — Adverse Event | 6
Not completed — Death | 11
Not completed — Insufficient clinical response | 1
Not completed — Withdrawal by Subject | 5
Not completed — Progressive disease | 2
Not completed — Other - Unspecified | 1

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) analysis set included all participants who received at least 1 of IV study medication during study.
Arm/Group | Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Parent Study (A4091003 [NCT00545129]) Baseline in Brief Pain Inventory-Short Form (BPI-sf) Average Pain Score for at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. It consists of 5 questions. Questions 1 to 4 measure the magnitude of pain at its worst, least, average, and 'right now'. Responses are provided by the participant on an 11 point numeric rating scale with anchors at 0 (No Pain) and 10 (Pain as bad as you can imagine). Measure can be scored by item, with lower scores being indicative of less pain. Negative Score indicates decrease in pain and Positive Score indicates increase in pain. This measure denotes the average pain score, minimum score = 0 and maximum score = 10 with lower scores indicative of less pain.
Time Frame: Baseline of Study A4091003, Baseline (A4091029) and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: The Intent to Treat (ITT) Population: all participants who received at least day 1 dose of IV study medication during Study A4091029. Here 'overall number of participants analyzed signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable at each specified category of specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029): Participants who received placebo in Study A4091003, were enrolled to Study A4091029 and received a single IV infusion of tanezumab 10 mg administered at Visit 1 (Baseline, Day 1), Visit 4 (Day 57, Week 8), Visit 6 (Day 113, Week 16), and Visit 7 (Day 169, Week 24). Participants in Poland entering the Extended-Use Period, tanezumab 10 mg was also administered via IV infusion at Visit 9 (Day 282, Week 40), Visit 10 (Day 337, Week 48), Visit 11 (Day 393, Week 56), and Visit 12 (Day 449, Week 64) with a plus or minus 5 day window for each post-baseline IV infusion.
- Tanezumab 10 mg (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029): Participants who received tanezumab 10 mg in Study A4091003, were enrolled to Study A4091029 and received a single IV infusion of tanezumab 10 mg administered at Visit 1 (Baseline, Day 1), Visit 4 (Day 57, Week 8), Visit 6 (Day 113, Week 16), and Visit 7 (Day 169, Week 24). Participants in Poland entering the Extended-Use Period, tanezumab 10 mg was also administered via IV infusion at Visit 9 (Day 282, Week 40), Visit 10 (Day 337, Week 48), Visit 11 (Day 393, Week 56), and Visit 12 (Day 449, Week 64) with a plus or minus 5 day window for each post-baseline IV infusion.
Arm/Group | Placebo (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029) | Tanezumab 10 mg (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline (A4091029) | -1.00 (2.16) | -1.17 (1.72)
  Week 4: number analyzed (Participants) | 18 | 17
  Week 4 | -1.67 (2.17) | -1.88 (1.76)
  Week 8: number analyzed (Participants) | 15 | 15
  Week 8 | -1.33 (1.50) | -1.87 (1.55)
  Week 16: number analyzed (Participants) | 12 | 13
  Week 16 | -1.58 (2.02) | -2.15 (2.41)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -1.60 (1.58) | -2.58 (1.68)
  Week 40: number analyzed (Participants) | 6 | 9
  Week 40 | 0.50 (1.38) | -2.44 (2.65)
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | -1.00
  Week 56: number analyzed (Participants) | 0 | 1
  Week 56 |  | -1.00
  Week 64: number analyzed (Participants) | 0 | 1
  Week 64 |  | -4.00

2. Primary Outcome: Change From A4091029 Baseline in BPI-sf Average Pain Score at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: as for outcome 1
Time Frame: Baseline and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: ITT Population. Here 'overall number of participants analyzed signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable at each specified category of specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 33
units on a scale
  Week 4 (n=33) | -0.82 (1.55)
  Week 8 (n=29): number analyzed (Participants) | 29
  Week 8 (n=29) | -0.69 (1.28)
  Week 16 (n=24): number analyzed (Participants) | 24
  Week 16 (n=24) | -0.67 (2.14)
  Week 24 (n=21): number analyzed (Participants) | 21
  Week 24 (n=21) | -1.19 (1.75)
  Week 40 (n=14): number analyzed (Participants) | 14
  Week 40 (n=14) | -0.21 (2.86)
  Week 48 (n=1): number analyzed (Participants) | 1
  Week 48 (n=1) | 0.00
  Week 56 (n=1): number analyzed (Participants) | 1
  Week 56 (n=1) | 0.00
  Week 64 (n=1): number analyzed (Participants) | 1
  Week 64 (n=1) | -3.00

3. Primary Outcome: Change From Parent Study (A4091003 [NCT00545129]) Baseline in BPI-sf Worst Pain Score at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. It consists of 5 questions. Questions 1 to 4 measure the magnitude of pain at its worst, least, average, and 'right now'. Responses are provided by the participant on an 11 point numeric rating scale with anchors at 0 (No Pain) and 10 (Pain as bad as you can imagine). Measure can be scored by item, with lower scores being indicative of less pain. Negative Score indicates decrease in pain and Positive Score indicates increase in pain. This measure denotes the worst pain score (within the last 24 hours at the time of the questionnaire), minimum score = 0 and maximum score = 10 with lower scores indicative of less pain.
Time Frame: Baseline of Study A4091003, Baseline (A4091029) and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029) | Tanezumab 10 mg (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline (A4091029) | -0.68 (2.69) | -0.72 (2.08)
  Week 4: number analyzed (Participants) | 18 | 17
  Week 4 | -1.22 (2.44) | -1.24 (1.71)
  Week 8: number analyzed (Participants) | 15 | 15
  Week 8 | -0.87 (2.17) | -0.87 (1.92)
  Week 16: number analyzed (Participants) | 12 | 13
  Week 16 | -0.67 (2.96) | -1.23 (2.68)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -1.20 (2.10) | -2.17 (1.99)
  Week 40: number analyzed (Participants) | 6 | 9
  Week 40 | -0.33 (2.07) | -2.11 (2.62)
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | -2.0
  Week 56: number analyzed (Participants) | 0 | 1
  Week 56 |  | -2.0
  Week 64: number analyzed (Participants) | 0 | 1
  Week 64 |  | -5.0

4. Primary Outcome: Change From Study A4091029 Baseline in BPI-sf Worst Pain Score at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: as for outcome 3
Time Frame: Baseline and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 33
units on a scale
  Week 4 | -0.82 (1.83)
  Week 8: number analyzed (Participants) | 29
  Week 8 | -0.48 (1.72)
  Week 16: number analyzed (Participants) | 24
  Week 16 | -0.25 (2.92)
  Week 24: number analyzed (Participants) | 21
  Week 24 | -1.14 (2.20)
  Week 40: number analyzed (Participants) | 14
  Week 40 | -0.36 (2.87)
  Week 48: number analyzed (Participants) | 1
  Week 48 | 0.00
  Week 56: number analyzed (Participants) | 1
  Week 56 | 0.00
  Week 64: number analyzed (Participants) | 1
  Week 64 | -3.00

5. Primary Outcome: Change From Parent Study (A4091003 [NCT00545129]) Baseline in BPI-sf Least Pain Score at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. It consists of 5 questions. Questions 1 to 4 measure the magnitude of pain at its worst, least, average, and 'right now'. Responses are provided by the participant on an 11 point numeric rating scale with anchors at 0 (No Pain) and 10 (Pain as bad as you can imagine). Measure can be scored by item, with lower scores being indicative of less pain. Negative Score indicates decrease in pain and Positive Score indicates increase in pain. This measure denotes the least pain score (within the last 24 hours at the time of the questionnaire), minimum score = 0 and maximum score = 10 with lower scores indicative of less pain.
Time Frame: Baseline of Study A4091003, Baseline (A4091029), and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029) | Tanezumab 10 mg (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline (A4091029) | -1.05 (2.04) | -1.28 (2.14)
  Week 4: number analyzed (Participants) | 18 | 17
  Week 4 | -2.28 (1.96) | -2.18 (2.07)
  Week 8: number analyzed (Participants) | 15 | 15
  Week 8 | -1.40 (1.76) | -2.60 (1.64)
  Week 16: number analyzed (Participants) | 12 | 13
  Week 16 | -1.67 (2.53) | -3.31 (2.32)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -2.50 (1.84) | -3.25 (1.82)
  Week 40: number analyzed (Participants) | 6 | 9
  Week 40 | -1.00 (1.67) | -2.67 (2.83)
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | -3.0
  Week 56: number analyzed (Participants) | 0 | 1
  Week 56 |  | -3.0
  Week 64: number analyzed (Participants) | 0 | 1
  Week 64 |  | -3.0

6. Primary Outcome: Change From Study A4091029 Baseline in BPI-sf Least Pain Score at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: as for outcome 5
Time Frame: Baseline and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 33
units on a scale
  Week 4 | -1.15 (1.46)
  Week 8: number analyzed (Participants) | 29
  Week 8 | -1.00 (1.36)
  Week 16: number analyzed (Participants) | 24
  Week 16 | -1.08 (1.93)
  Week 24: number analyzed (Participants) | 21
  Week 24 | -1.81 (1.60)
  Week 40: number analyzed (Participants) | 14
  Week 40 | -1.00 (2.11)
  Week 48: number analyzed (Participants) | 1
  Week 48 | -1.00
  Week 56: number analyzed (Participants) | 1
  Week 56 | -1.00
  Week 64: number analyzed (Participants) | 1
  Week 64 | -1.00

7. Primary Outcome: Change From Parent Study (A4091003 [NCT00545129]) Baseline in BPI-sf Score for Right Now Pain at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. It consists of 5 questions. Questions 1 to 4 measure the magnitude of pain at its worst, least, average, and 'right now'. Responses are provided by the participant on an 11 point numeric rating scale with anchors at 0 (No Pain) and 10 (Pain as bad as you can imagine). Measure can be scored by item, with lower scores being indicative of less pain. Negative Score indicates decrease in pain and Positive Score indicates increase in pain. This measure denotes the right now pain score (at the time of the questionnaire), minimum score = 0 and maximum score = 10 with lower scores indicative of less pain.
Time Frame: Baseline of Study A4091003, Baseline (A4091029), and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029) | Tanezumab 10 mg (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline (A4091029) | -0.68 (2.73) | -1.61 (1.85)
  Week 4: number analyzed (Participants) | 18 | 17
  Week 4 | -1.67 (1.94) | -2.24 (2.31)
  Week 8: number analyzed (Participants) | 15 | 15
  Week 8 | -1.20 (1.82) | -2.40 (2.16)
  Week 16: number analyzed (Participants) | 12 | 13
  Week 16 | -1.08 (2.64) | -2.54 (3.04)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -1.20 (1.48) | -2.75 (2.56)
  Week 40: number analyzed (Participants) | 6 | 9
  Week 40 | 0.00 (1.10) | -2.11 (3.76)
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | -2.00
  Week 56: number analyzed (Participants) | 0 | 1
  Week 56 |  | -4.00
  Week 64: number analyzed (Participants) | 0 | 1
  Week 64 |  | -4.00

8. Primary Outcome: Change From Study A4091029 Baseline in BPI-sf Score for Right Now Pain at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: as for outcome 7
Time Frame: Baseline and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 33
units on a scale
  Week 4 | -0.82 (1.61)
  Week 8: number analyzed (Participants) | 29
  Week 8 | -0.72 (1.62)
  Week 16: number analyzed (Participants) | 24
  Week 16 | -0.67 (2.62)
  Week 24: number analyzed (Participants) | 21
  Week 24 | -0.95 (1.72)
  Week 40: number analyzed (Participants) | 14
  Week 40 | -0.21 (3.49)
  Week 48: number analyzed (Participants) | 1
  Week 48 | -1.00
  Week 56: number analyzed (Participants) | 1
  Week 56 | -3.00
  Week 64: number analyzed (Participants) | 1
  Week 64 | -3.00

9. Primary Outcome: Change From Parent Study (A4091003 [NCT00545129]) Baseline in BPI-sf Score for Pain Interference With Function (Composite Score) Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. It consists of 5 questions. Question 5 consists of seven item subsets, A to G, that measure the level of interference of pain on daily functions. Responses are given on an 11 point numeric rating scale with anchors at 0 (Does not interfere) and 10 (Completely interferes). Measure can be scored by item, with lower scores being indicative of less pain interference. The BPI-sf Pain Interference with Function Composite score is calculated as the average of the seven item subsets (questions 5A to G) in the BPI-sf questionnaire. If one of the seven items was missing then the average score of the remaining items was used to impute the missing (seventh) value. If more than one item was missing then the composite score was missing.
Time Frame: Baseline of Study A4091003, Baseline (A4091029), and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029) | Tanezumab 10 mg (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline (A4091029) | -0.81 (2.32) | -1.10 (2.11)
  Week 4: number analyzed (Participants) | 17 | 17
  Week 4 | -2.03 (2.02) | -1.26 (1.91)
  Week 8: number analyzed (Participants) | 14 | 15
  Week 8 | -1.22 (1.49) | -1.61 (2.13)
  Week 16: number analyzed (Participants) | 11 | 13
  Week 16 | -1.05 (2.35) | -1.38 (2.56)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -1.41 (1.84) | -1.94 (1.87)
  Week 40: number analyzed (Participants) | 6 | 8
  Week 40 | -0.90 (2.04) | -2.38 (2.89)
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | -3.00
  Week 56: number analyzed (Participants) | 0 | 1
  Week 56 |  | -3.29
  Week 64: number analyzed (Participants) | 0 | 1
  Week 64 |  | -5.43

10. Primary Outcome: Change From Study A4091029 Baseline in BPI-sf Score for Pain Interference With Function (Composite Score) at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: as for outcome 9
Time Frame: Baseline and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 33
units on a scale
  Week 4 | -0.69 (1.33)
  Week 8: number analyzed (Participants) | 29
  Week 8 | -0.79 (1.90)
  Week 16: number analyzed (Participants) | 24
  Week 16 | -0.29 (2.46)
  Week 24: number analyzed (Participants) | 21
  Week 24 | -0.88 (1.77)
  Week 40: number analyzed (Participants) | 13
  Week 40 | -0.56 (2.81)
  Week 48: number analyzed (Participants) | 1
  Week 48 | -1.71
  Week 56: number analyzed (Participants) | 1
  Week 56 | -2.00
  Week 64: number analyzed (Participants) | 1
  Week 64 | -4.14

11. Primary Outcome: Change From Parent Study (A4091003 [NCT00545129]) Baseline in BPI-sf Item Scores for Pain Interference at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. It consists of 5 questions. Question 5 consists of seven item subsets, A to G, that measure the level of interference of pain on daily functions. Items are defined as interference with, general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life mood. Responses are given on an 11 point numeric rating scale with anchors at 0 (Does not interfere) and 10 (Completely interferes). Measure can be scored by item, with lower scores being indicative of less pain interference.
Time Frame: Baseline of Study A4091003, Baseline (A4091029), and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029) | Tanezumab 10 mg (A4091003 [NCT00545129]) to Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 19 | 18
units on a scale
  General activity: Baseline | -0.68 (2.65) | -1.39 (2.57)
  General activity: Week 4: number analyzed (Participants) | 18 | 17
  General activity: Week 4 | -1.94 (2.04) | -1.76 (2.11)
  General activity: Week 8: number analyzed (Participants) | 15 | 15
  General activity: Week 8 | -1.47 (2.17) | -2.27 (2.19)
  General activity: Week 16: number analyzed (Participants) | 12 | 13
  General activity: Week 16 | -1.00 (2.95) | -1.31 (3.09)
  General activity: Week 24: number analyzed (Participants) | 10 | 12
  General activity: Week 24 | -1.60 (1.71) | -2.17 (2.37)
  General activity: Week 40: number analyzed (Participants) | 6 | 9
  General activity: Week 40 | -0.83 (1.72) | -2.78 (3.03)
  General activity: Week 48: number analyzed (Participants) | 0 | 1
  General activity: Week 48 |  | -3.00
  General activity: Week 56: number analyzed (Participants) | 0 | 1
  General activity: Week 56 |  | -3.00
  General activity: Week 64: number analyzed (Participants) | 0 | 1
  General activity: Week 64 |  | -6.00
  Mood: Baseline | -1.58 (1.98) | -0.94 (2.78)
  Mood: Week 4: number analyzed (Participants) | 18 | 17
  Mood: Week 4 | -2.33 (1.78) | -1.53 (2.48)
  Mood: Week 8: number analyzed (Participants) | 15 | 15
  Mood: Week 8 | -2.27 (2.43) | -1.53 (2.72)
  Mood: Week 16: number analyzed (Participants) | 12 | 13
  Mood: Week 16 | -1.50 (2.97) | -1.62 (3.57)
  Mood: Week 24: number analyzed (Participants) | 10 | 12
  Mood: Week 24 | -2.20 (2.90) | -1.58 (2.87)
  Mood: Week 40: number analyzed (Participants) | 6 | 9
  Mood: Week 40 | -1.00 (2.97) | -2.56 (3.05)
  Mood: Week 48: number analyzed (Participants) | 0 | 1
  Mood: Week 48 |  | -4.00
  Mood: Week 56: number analyzed (Participants) | 0 | 1
  Mood: Week 56 |  | -4.00
  Mood: Week 64: number analyzed (Participants) | 0 | 1
  Mood: Week 64 |  | -7.00
  Walking ability: Baseline: number analyzed (Participants) | 18 | 18
  Walking ability: Baseline | -0.67 (2.77) | -0.17 (2.57)
  Walking ability: Week 4: number analyzed (Participants) | 17 | 17
  Walking ability: Week 4 | -1.65 (2.57) | -0.24 (2.25)
  Walking ability: Week 8: number analyzed (Participants) | 14 | 15
  Walking ability: Week 8 | -0.86 (2.25) | -0.73 (1.83)
  Walking ability: Week 16: number analyzed (Participants) | 11 | 13
  Walking ability: Week 16 | -1.00 (2.93) | -0.23 (1.88)
  Walking ability: Week 24: number analyzed (Participants) | 10 | 12
  Walking ability: Week 24 | -1.00 (2.75) | -0.92 (1.88)
  Walking ability: Week 40: number analyzed (Participants) | 6 | 8
  Walking ability: Week 40 | -1.50 (2.81) | -0.63 (3.07)
  Walking ability: Week 48: number analyzed (Participants) | 0 | 1
  Walking ability: Week 48 |  | -3.00
  Walking ability: Week 56: number analyzed (Participants) | 0 | 1
  Walking ability: Week 56 |  | -4.00
  Walking ability: Week 64: number analyzed (Participants) | 0 | 1
  Walking ability: Week 64 |  | -5.00
  Normal work: Baseline: number analyzed (Participants) | 18 | 18
  Normal work: Baseline | -0.28 (2.85) | -1.28 (2.61)
  Normal work: Week 4: number analyzed (Participants) | 17 | 17
  Normal work: Week 4 | -1.41 (3.43) | -1.12 (2.74)
  Normal work: Week 8: number analyzed (Participants) | 14 | 15
  Normal work: Week 8 | -0.50 (2.71) | -1.93 (2.94)
  Normal work: Week 16: number analyzed (Participants) | 11 | 13
  Normal work: Week 16 | -1.00 (2.28) | -1.00 (3.29)
  Normal work: Week 24: number analyzed (Participants) | 10 | 12
  Normal work: Week 24 | -1.10 (2.33) | -1.75 (2.83)
  Normal work: Week 40: number analyzed (Participants) | 6 | 8
  Normal work: Week 40 | -0.67 (2.88) | -1.88 (4.49)
  Normal work: Week 48: number analyzed (Participants) | 0 | 1
  Normal work: Week 48 |  | 1.00
  Normal work: Week 56: number analyzed (Participants) | 0 | 1
  Normal work: Week 56 |  | 0.00
  Normal work: Week 64: number analyzed (Participants) | 0 | 1
  Normal work: Week 64 |  | -3.00
  Relations with other people: Baseline: number analyzed (Participants) | 18 | 18
  Relations with other people: Baseline | -0.50 (2.92) | -1.28 (2.44)
  Relations with other people: Week 4: number analyzed (Participants) | 17 | 17
  Relations with other people: Week 4 | -2.41 (2.50) | -1.41 (2.29)
  Relations with other people: Week 8: number analyzed (Participants) | 14 | 15
  Relations with other people: Week 8 | -1.00 (2.04) | -1.47 (2.64)
  Relations with other people: Week 16: number analyzed (Participants) | 11 | 13
  Relations with other people: Week 16 | -1.36 (3.20) | -1.31 (2.50)
  Relations with other people: Week 24: number analyzed (Participants) | 10 | 12
  Relations with other people: Week 24 | -1.40 (2.99) | -1.92 (2.31)
  Relations with other people: Week 40: number analyzed (Participants) | 6 | 9
  Relations with other people: Week 40 | -1.17 (2.23) | -1.89 (3.06)
  Relations with other people: Week 48: number analyzed (Participants) | 0 | 1
  Relations with other people: Week 48 |  | -3.00
  Relations with other people: Week 56: number analyzed (Participants) | 0 | 1
  Relations with other people: Week 56 |  | -3.00
  Relations with other people: Week 64: number analyzed (Participants) | 0 | 1
  Relations with other people: Week 64 |  | -5.00
  Sleep: Baseline: number analyzed (Participants) | 18 | 18
  Sleep: Baseline | -1.00 (2.89) | -1.00 (2.43)
  Sleep: Week 4: number analyzed (Participants) | 17 | 17
  Sleep: Week 4 | -2.18 (2.32) | -1.59 (2.53)
  Sleep: Week 8: number analyzed (Participants) | 14 | 15
  Sleep: Week 8 | -1.21 (2.01) | -1.47 (3.16)
  Sleep: Week 16: number analyzed (Participants) | 11 | 13
  Sleep: Week 16 | -1.09 (1.81) | -1.85 (3.02)
  Sleep: Week 24: number analyzed (Participants) | 10 | 12
  Sleep: Week 24 | -0.60 (1.90) | -2.08 (2.75)
  Sleep: Week 40: number analyzed (Participants) | 6 | 9
  Sleep: Week 40 | -0.17 (1.83) | -3.11 (3.18)
  Sleep: Week 48: number analyzed (Participants) | 0 | 1
  Sleep: Week 48 |  | -5.00
  Sleep: Week 56: number analyzed (Participants) | 0 | 1
  Sleep: Week 56 |  | -5.00
  Sleep: Week 64: number analyzed (Participants) | 0 | 1
  Sleep: Week 64 |  | -5.00
  Enjoyment of life: Baseline: number analyzed (Participants) | 18 | 18
  Enjoyment of life: Baseline | -1.39 (2.99) | -1.67 (2.72)
  Enjoyment of life: Week 4: number analyzed (Participants) | 17 | 17
  Enjoyment of life: Week 4 | -2.53 (2.92) | -1.18 (2.77)
  Enjoyment of life: Week 8: number analyzed (Participants) | 14 | 15
  Enjoyment of life: Week 8 | -1.71 (2.64) | -1.87 (3.38)
  Enjoyment of life: Week 16: number analyzed (Participants) | 11 | 13
  Enjoyment of life: Week 16 | -1.09 (2.43) | -2.38 (3.50)
  Enjoyment of life: Week 24: number analyzed (Participants) | 10 | 12
  Enjoyment of life: Week 24 | -2.00 (2.36) | -3.17 (2.12)
  Enjoyment of life: Week 40: number analyzed (Participants) | 6 | 8
  Enjoyment of life: Week 40 | -1.00 (3.58) | -3.38 (3.46)
  Enjoyment of life: Week 48: number analyzed (Participants) | 0 | 1
  Enjoyment of life: Week 48 |  | -4.00
  Enjoyment of life: Week 56: number analyzed (Participants) | 0 | 1
  Enjoyment of life: Week 56 |  | -4.00
  Enjoyment of life: Week 64: number analyzed (Participants) | 0 | 1
  Enjoyment of life: Week 64 |  | -7.00

12. Primary Outcome: Change From Study A4091029 Baseline in BPI-sf Item Scores for Pain Interference at Weeks 4, 8, 16, 24, 40, 48, 56 and 64
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. It consists of 5 questions. Question 5 consists of seven item subsets, A to G, that measure the level of interference of pain on daily functions. Items are defined as interference with: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life mood. Responses are given on an 11 point numeric rating scale with anchors at 0 (Does not interfere) and 10 (Completely interferes). Measure can be scored by item, with lower scores being indicative of less pain interference.
Time Frame: Baseline and Weeks 4, 8, 16, 24, 40, 48, 56 and 64 of Study A4091029
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mg (A4091029)
Number analyzed (Participants) | 33
units on a scale
  General activity: Week 4 | -0.85 (1.84)
  General activity: Week 8: number analyzed (Participants) | 29
  General activity: Week 8 | -1.10 (2.27)
  General activity: Week 16: number analyzed (Participants) | 24
  General activity: Week 16 | 0.04 (2.90)
  General activity: Week 24: number analyzed (Participants) | 21
  General activity: Week 24 | -0.90 (2.32)
  General activity: Week 40: number analyzed (Participants) | 14
  General activity: Week 40 | -0.57 (2.93)
  General activity: Week 48: number analyzed (Participants) | 1
  General activity: Week 48 | -1.00
  General activity: Week 56: number analyzed (Participants) | 1
  General activity: Week 56 | -1.00
  General activity: Week 64: number analyzed (Participants) | 1
  General activity: Week 64 | -4.00
  Mood: Week 4 | -0.70 (1.55)
  Mood: Week 8: number analyzed (Participants) | 29
  Mood: Week 8 | -0.86 (2.26)
  Mood: Week 16: number analyzed (Participants) | 24
  Mood: Week 16 | -0.21 (2.77)
  Mood: Week 24: number analyzed (Participants) | 21
  Mood: Week 24 | -0.62 (1.88)
  Mood: Week 40: number analyzed (Participants) | 14
  Mood: Week 40 | -0.14 (3.13)
  Mood: Week 48: number analyzed (Participants) | 1
  Mood: Week 48 | -2.00
  Mood: Week 56: number analyzed (Participants) | 1
  Mood: Week 56 | -2.00
  Mood: Week 64: number analyzed (Participants) | 1
  Mood: Week 64 | -5.00
  Walking ability: Week 4 ( | -0.61 (1.60)
  Walking ability: Week 8: number analyzed (Participants) | 29
  Walking ability: Week 8 | -0.79 (1.90)
  Walking ability: Week 16: number analyzed (Participants) | 24
  Walking ability: Week 16 | -0.50 (2.11)
  Walking ability: Week 24: number analyzed (Participants) | 21
  Walking ability: Week 24 | -1.05 (2.06)
  Walking ability: Week 40: number analyzed (Participants) | 13
  Walking ability: Week 40 | -1.08 (2.90)
  Walking ability: Week 48: number analyzed (Participants) | 1
  Walking ability: Week 48 | -2.00
  Walking ability: Week 56: number analyzed (Participants) | 1
  Walking ability: Week 56 | -3.00
  Walking ability: Week 64: number analyzed (Participants) | 1
  Walking ability: Week 64 | -4.00
  Normal work: Week 4 | -0.42 (2.02)
  Normal work: Week 8: number analyzed (Participants) | 29
  Normal work: Week 8 | -0.62 (2.41)
  Normal work: Week 16: number analyzed (Participants) | 24
  Normal work: Week 16 | 0.08 (2.78)
  Normal work: Week 24: number analyzed (Participants) | 21
  Normal work: Week 24 | -0.76 (1.87)
  Normal work: Week 40: number analyzed (Participants) | 13
  Normal work: Week 40 | -0.46 (3.36)
  Normal work: Week 48: number analyzed (Participants) | 1
  Normal work: Week 48 | -1.00
  Normal work: Week 56: number analyzed (Participants) | 1
  Normal work: Week 56 | -2.00
  Normal Work: Week 64: number analyzed (Participants) | 1
  Normal Work: Week 64 | -5.00
  Relations with other people: Week 4 | -1.18 (2.05)
  Relations with other people: Week 8: number analyzed (Participants) | 29
  Relations with other people: Week 8 | -0.86 (2.43)
  Relations with other people: Week 16: number analyzed (Participants) | 24
  Relations with other people: Week 16 | -0.67 (2.46)
  Relations with other people: Week 24: number analyzed (Participants) | 21
  Relations with other people: Week 24 | -1.19 (2.09)
  Relations with other people: Week 40: number analyzed (Participants) | 14
  Relations with other people: Week 40 | -0.71 (2.70)
  Relations with other people: Week 48: number analyzed (Participants) | 1
  Relations with other people: Week 48 | -3.00
  Relations with other people: Week 56: number analyzed (Participants) | 1
  Relations with other people: Week 56 | -3.00
  Relations with other people: Week 64: number analyzed (Participants) | 1
  Relations with other people: Week 64 | -5.00
  Sleep: Week 4 | -0.94 (1.60)
  Sleep: Week 8: number analyzed (Participants) | 29
  Sleep: Week 8 | -0.76 (2.15)
  Sleep: Week 16: number analyzed (Participants) | 24
  Sleep: Week 16 | -0.63 (2.73)
  Sleep: Week 24: number analyzed (Participants) | 21
  Sleep: Week 24 | -0.86 (2.20)
  Sleep: Week 40: number analyzed (Participants) | 14
  Sleep: Week 40 | -0.71 (2.76)
  Sleep: Week 48: number analyzed (Participants) | 1
  Sleep: Week 48 | -1.00
  Sleep: Week 56: number analyzed (Participants) | 1
  Sleep: Week 56 | -1.00
  Sleep: Week 64: number analyzed (Participants) | 1
  Sleep: Week 64 | -1.00
  Enjoyment of life: Week 4 | -0.12 (1.75)
  Enjoyment of life: Week 8: number analyzed (Participants) | 29
  Enjoyment of life: Week 8 | -0.55 (2.57)
  Enjoyment of life: Week 16: number analyzed (Participants) | 24
  Enjoyment of life: Week 16 | -0.17 (3.12)
  Enjoyment of life: Week 24: number analyzed (Participants) | 21
  Enjoyment of life: Week 24 | -0.81 (2.40)
  Enjoyment of life: Week 40: number analyzed (Participants) | 13
  Enjoyment of life: Week 40 | -0.08 (3.75)
  Enjoyment of life: Week 48: number analyzed (Participants) | 1
  Enjoyment of life: Week 48 | -2.00
  Enjoyment of life: Week 56: number analyzed (Participants) | 1
  Enjoyment of life: Week 56 | -2.00
  Enjoyment of life: Week 64: number analyzed (Participants) | 1
  Enjoyment of life: Week 64 | -5.00

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Tanezumab 10 mg (A4091029)
Serious Adverse Events (participants affected / at risk) | 23/41
Other Adverse Events (participants affected / at risk) | 18/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 10 mg (A4091029) (N=41)
Anaemia (Blood and lymphatic system disorders) | 4
Aplastic anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disease progression (General disorders) | 3
Cardiovascular insufficiency (Cardiac disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Renal failure acute (Renal and urinary disorders) | 1
Hepatorenal failure (Hepatobiliary disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 10 mg (A4091029) (N=41)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 6
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 5
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less